CLINICAL TRIAL: NCT01259310
Title: Women With Epilepsy: Pregnancy Outcomes and Deliveries
Acronym: WEPOD
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Brigham and Women's Hospital (Other); Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: WEPOD
Record Dates: First submitted 2010-12-10; First posted 2010-12-14 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Epilepsy
Keywords: fertility; women; epilepsy; pregnancy; seizures; seizure frequency; ovulation; menstruation; hormones; progesterone
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Women with epilepsy: Women with epilepsy, age 18-40 years, who express a desire to conceive and have stopped or plan to stop taking birth control.
- Women without epilepsy: Healthy women, age 18-40 years, who express a desire to conceive and have stopped or plan to stop taking birth control.

SUMMARY:
This is a three-center prospective case-control study to examine the patterns of fertility among women with epilepsy (WWE) compared to an age-matched group of women without epilepsy (WWoE).

DETAILED DESCRIPTION:
This is a three-center prospective case-control study to examine the patterns of fertility among women with epilepsy (WWE) compared to an age-matched group of women without epilepsy (WWoE). The investigators will determine if pregnancy rates differ in WWE compared to WWoE. Covariates of interest include proportion of ovulatory cycles, sexual activity, and type of anti-epileptic drug (AED). The investigators will compare seizure frequency during preconception to seizure frequency during pregnancy, with analysis of covariates of interest (AED type, AED ratio-to-target concentrations, and epilepsy syndrome). The investigators will also observe interactions between seizures/epilepsy, AEDs, and sex steroid hormones during this opportune time when women are not on birth control. Patterns of seizures will be evaluated for accepted catamenial patterns with consideration of ovulatory and anovulatory cycles, AED concentrations, and epilepsy type.

ELIGIBILITY:
Inclusion Criteria:

* between ages 18 and 40
* planning pregnancy
* stopped birth control or planning to stop birth control
* for women with epilepsy: receiving at least one AED (lamotrigine, levetiracetam, carbamazepine, phenytoin, oxcarbazepine, phenobarbital, topiramate, rufinamide). If on polytherapy, AEDs cannot include lamotrigine, levetiracetam or valproate.

Exclusion Criteria:

* Use of hormonal therapies for contraception
* demonstrated infertility with the same partner (more than 12 months of unprotected intercourse without achieving pregnancy)
* diagnosis of infertility
* Polycystic ovarian syndrome
* severe endometriosis
* currently breastfeeding
* male factor infertility
* surgical or medical menopause
* smokers who have more than 10 cigarettes per day
* untreated thyroid disease
* hyperprolactinemia or other pituitary disease
* recently trying to achieve pregnancy for more than 6 months with having regular vaginal sexual intercourse without contraception

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with epilepsy between 18 and 40 years of age, recruited from epilepsy clinics in New York and Boston, and control women without epilepsy between 18 and 40 years of age, recruited from Obstetrics and Gynaecology clinics, local academic institutions, and referrals from epilepsy clinic employees or patients.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2010-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Fertility in women with epilepsy compared to healthy controls | 1.75 years
  Percentage of women who have a live birth within the time frame.

SECONDARY OUTCOMES:
Seizure frequency in women with epilepsy at baseline compared to during pregnancy | 1.75 years

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline French, MD, Principal Investigator — NYU School of Medicine; Page Pennell, MD, Principal Investigator — Brigham and Women's Hospital; Cynthia Harden, MD, Principal Investigator — Northwell Health
Locations (3):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - North Shore Long Island Jewish Health System, Great Neck, New York
  - NYU Langone Medical Center, New York, New York